CLINICAL TRIAL: NCT01221285
Title: A Biomarker-Based Pilot Study of Cockroach Subcutaneous Immunotherapy in Cockroach Sensitive Adults With Asthma and/or Perennial Allergic Rhinitis (ICAC-18)
Brief Title: Development of Cockroach Immunotherapy by the Inner-City Asthma Consortium
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Inner-City Asthma Consortium (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DAIT ICAC-18; SCITCO (Other: NIAID)
Record Dates: First submitted 2010-10-13; First posted 2010-10-14 (Estimated); Results first posted 2014-05-23 (Estimated); Last update posted 2014-06-11 (Estimated); Status verified 2014-06

CONDITIONS: Asthma; Perennial Allergic Rhinitis
Keywords: Cockroach; Immunotherapy; Subcutaneous immunotherapy; Inner city asthma
MeSH Terms: conditions — Asthma; Rhinitis, Allergic, Perennial

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- German cockroach allergenic extract (Experimental): Participants will receive weekly escalating doses of glycerinated German cockroach allergenic extract administered via the subcutaneous route up to a Maximum Study Dose of 0.6 mL of extract at a concentration of 1:20 wt/vol.
  Interventions: Biological: German cockroach (Blattella germanica) allergenic extract

INTERVENTIONS:
Biological: German cockroach (Blattella germanica) allergenic extract — Participants received weekly escalating doses of glycerinated German cockroach allergenic extract administered via the subcutaneous route up to a Maximum Study Dose of 0.6 mL of extract at a concentration of 1:20 wt/vol.

SUMMARY:
This trial is a biomarker-based pilot study of the safety of Cockroach Subcutaneous Immunotherapy in Cockroach-sensitive Adults (SCITCO) who have a history of perennial allergic rhinitis, asthma, or both.

DETAILED DESCRIPTION:
Scientific evidence has shown that, over the past two decades, the combination of cockroach allergy and cockroach exposure is one of the most important factors contributing to the dramatic increase in asthma morbidity seen in inner city children with asthma. Therefore, a major goal of the Inner City Asthma Consortium (ICAC) is to evaluate the efficacy of cockroach immunotherapy in inner city asthma.

ELIGIBILITY:
Inclusion Criteria:

* Have a history of perennial allergic rhinitis, asthma, or both, for a minimum of 1 year before study entry. For those with asthma:

  * a diagnosis of asthma will be defined as a report by the participant that they have had a clinical diagnosis of asthma made by a physician over a year ago
  * the participant's asthma must be well controlled as defined by:
  * a forced expiratory volume at one second (FEV1) greater than or equal to 80% predicted value with or without controller medication
  * albuterol use for no more than 3 days per week in each of the previous 2 weeks for asthma symptoms (not including exercise prophylaxis)
* Are sensitive to German cockroach (Blattella germanica) as documented by a positive (>= 3 mm greater than negative control) skin prick test result and detectable German cockroach specific IgE (>=0.35 kUA/L)
* Have no known contraindications to therapy with glycerinated German (Blattella germanica) cockroach allergenic extract
* Are willing to sign the written Informed Consent prior to initiation of any study procedure

Exclusion Criteria:

* Are pregnant or lactating. Females must be abstinent or use a medically acceptable birth control method throughout the study (e.g. oral, subcutaneous, mechanical, or surgical contraception)
* Are unable to perform spirometry at screening
* Have an asthma severity classification at recruitment of severe persistent, using the National Asthma Education and Prevention Program (NAEPP) classification, as evidenced by at least one of the following:

  * requires a dose of greater than 500 mcg of fluticasone per day or the equivalent of another inhaled corticosteroid
  * have received more than 2 courses of oral or parenteral corticosteroids within the last 12 months
  * have been treated with depot steroids within the last 12 months
  * have been hospitalized for asthma within the 6 months prior to recruitment
  * have had a life-threatening asthma exacerbation that required intubation, mechanical ventilation, or that resulted in a hypoxic seizure within 2 years prior to recruitment
* Do not have access to a phone (needed for scheduling appointments)
* Have received allergen immunotherapy (SLIT or SCIT) in the last 12 months prior to recruitment or who plan to initiate or resume allergen immunotherapy during the study. Subjects who only received placebo therapy in the BioCSI protocol (A Biomarker-based Pilot Study of Cockroach Sublingual Immunotherapy in Cockroach Sensitive Adults With Asthma and/or Perennial Allergic Rhinitis, ICAC-12, NCT00829985) are eligible to participate in this study
* Have previously been treated with anti-IgE therapy within 1 year of recruitment
* Have received an investigational drug in the 30 days prior to recruitment or who plan to use an investigational drug during the study
* Refuse to sign the Epinephrine Auto-injector Training Form
* Do not primarily speak English
* Plan to move from the area during the study period
* Have a history of idiopathic anaphylaxis or anaphylaxis grade 2 or higher as defined in the protocol
* Have unstable angina, significant arrhythmia, uncontrolled hypertension, history of autoimmune disease, or other chronic or immunological diseases that in the opinion of the investigator might interfere with the evaluation of the investigational agent or pose additional risk to the participant
* Are using tricyclic antidepressants or beta-adrenergic blocker drugs (either oral or topical route[s] of administration)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2010-09; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Wood, MD, Study Chair — Johns Hopkins University
Locations (1):
- Johns Hopkins University School of Medicine, Baltimore, Maryland, United States

REFERENCES:
- [Result] Wood RA, Togias A, Wildfire J, Visness CM, Matsui EC, Gruchalla R, Hershey G, Liu AH, O'Connor GT, Pongracic JA, Zoratti E, Little F, Granada M, Kennedy S, Durham SR, Shamji MH, Busse WW. Development of cockroach immunotherapy by the Inner-City Asthma Consortium. J Allergy Clin Immunol. 2014 Mar;133(3):846-52.e6. doi: 10.1016/j.jaci.2013.08.047. Epub 2013 Nov 1. PMID 24184147

RESULTS

PARTICIPANT FLOW:
Groups:
- Glycerinated German Cockroach Allergenic Extract: Participants received weekly escalating doses of glycerinated German cockroach allergenic extract administered via the subcutaneous route up to a Maximum Study Dose of 0.6 ml of extract at a concentration of 1:20 wt/vol.
Period: Overall Study
Arm/Group | Glycerinated German Cockroach Allergenic Extract
Started | 11
Completed | 10
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Glycerinated German Cockroach Allergenic Extract
Number analyzed (Participants) | 10
Age, Continuous [Median (Full Range); unit: years] | 37.5 [24 to 52]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 10
Participants with Asthma [Number; unit: participants] — Participants who were diagnosed with asthma by a physician for a minimum of 1 year prior to study enrollment
  participants | 7
Participants with Perennial Allergic Rhinitis [Number; unit: participants] — Participants reporting sneezing, nasal congestion or runny nose symptoms greater or equal to 3 days per week for 4 or more months in the year preceding study enrollment
  participants | 6
Glycerinated German Cockroach Prick Skin Test Wheal Size [Median (Full Range); unit: mm] — German cockroach prick skin test wheal size at screening. A measurable wheal when exposed to cockroach allergen extract by prick skin test (as compared to the negative control wheal) is a sign of allergic sensitization ("allergy") to cockroach. Higher wheal sizes indicate greater allergic reaction or sensitization.
  mm | 6.8 [3 to 9]
German Cockroach-Specific Serum Immunoglobulin E (IgE) Levels [Median (Full Range); unit: kU/L] — German cockroach-specific serum IgE levels at screening.
  kU/L | 3.8 [0.9 to 24.9]

OUTCOME MEASURES:

1. Primary Outcome: Number of Reported Treatment-related Adverse Events (AEs)
Description: Number of non-serious adverse events reported as possibly related, probably related, or definitely related to study participation.
Time Frame: Baseline through 6-months of treatment
Population: Intent-to-treat
Measure: Number; unit: Events
Arm/Group | Glycerinated German Cockroach Allergenic Extract
Number analyzed (Participants) | 10
Events
  Severe, Definitely | 0
  Severe, Probably | 0
  Severe, Possibly | 0
  Moderate, Definitely | 0
  Moderate , Probably | 3
  Moderate , Possibly | 1
  Mild , Definitely | 0
  Mild Probably | 47
  Mild Possibly | 99

2. Primary Outcome: Number of Reported Treatment-related Serious Adverse Events (SAEs)
Description: Number of SAEs reported as possibly related, probably related, or definitely related to study participation.
Time Frame: Baseline through 6-months of treatment
Population: Intent-to-treat
Measure: Number; unit: Events
Arm/Group | Glycerinated German Cockroach Allergenic Extract
Number analyzed (Participants) | 10
Events
  Definitely related | 0
  Probably related | 0
  Possibly related | 0

3. Secondary Outcome: Change in German Cockroach-Specific Serum IgE Over Time
Description: Outcome is the ratio of geometric means for baseline German cockroach-specific serum Immunoglobulin E (IgE) vs. post-baseline German cockroach-specific serum IgE. Numerator is geometric mean post-baseline IgE; denominator is baseline IgE. This result is an indicator of immune modulation over time, however its clinical significance is unclear.
Time Frame: Baseline through 6-months of treatment
Population: Intent-to-treat
Measure: Number (95% Confidence Interval); unit: Ratio
Arm/Group | Glycerinated German Cockroach Allergenic Extract
Number analyzed (Participants) | 10
Ratio | 1.8 (0.1) [1.1 to 2.8]
Statistical Analysis 1: Comparison: Glycerinated German Cockroach Allergenic Extract; Test type: Superiority or Other; p = 0.02, Fold change; Fold change = 1.8, 95% CI 2-sided [1.1 to 2.8] — Numerator is geometric mean post-baseline IgE. Denominator is baseline IgE

4. Secondary Outcome: Change in German Cockroach-Specific Serum IgG Over Time
Description: Outcome is the ratio of geometric means for baseline German cockroach-specific serum Immunoglobulin G (IgG) vs. post-baseline German cockroach-specific serum IgG. Numerator is geometric mean post-baseline IgG; denominator is baseline IgG.This result is an indicator of immune modulation over time, however its clinical significance is unclear.
Time Frame: Baseline through 6-months of treatment
Population: Intent-to-treat
Measure: Number (95% Confidence Interval); unit: Ratio
Arm/Group | Glycerinated German Cockroach Allergenic Extract
Number analyzed (Participants) | 10
Ratio | 2.5 (0.1) [1.8 to 3.4]
Statistical Analysis 1: Comparison: Glycerinated German Cockroach Allergenic Extract; Test type: Superiority or Other; p < 0.0001, Fold change; Fold change = 2.5, 95% CI 2-sided [1.8 to 3.4] — Numerator is geometric mean post-baseline IgG. Denominator is baseline IgG

5. Secondary Outcome: Change in German Cockroach-Specific Serum IgG4 Over Time
Description: Outcome is the ratio of geometric means for baseline German cockroach-specific serum Immunoglobulin subclass 4 (IgG4) vs. post-baseline German cockroach-specific serum IgG4. Numerator is geometric mean post-baseline IgG4; denominator is baseline IgG4. This result is an indicator of immune modulation over time, however its clinical significance is unclear.
Time Frame: Baseline through 6-months of treatment
Population: Intent-to-treat
Measure: Number (95% Confidence Interval); unit: Ratio
Arm/Group | Glycerinated German Cockroach Allergenic Extract
Number analyzed (Participants) | 10
Ratio | 12.9 (0.7) [7.5 to 22.5]
Statistical Analysis 1: Comparison: Glycerinated German Cockroach Allergenic Extract; Test type: Superiority or Other; p < 0.0001, Fold Change; Fold change = 12.9, 95% CI 2-sided [7.5 to 22.5] — Numerator is geometric mean post-baseline IgG4. Denominator is baseline IgG4

6. Secondary Outcome: Change in IgE Fragment Antibody Binding (FAB) Activity (10 Micrograms/mL Cockroach Allergen Extract)
Description: Outcome is the change in mean IgE fragment antibody binding (FAB) activity, baseline to post-baseline. Serum from cockroach subcutaneous immunotherapy (SCIT)-treated participants were analyzed to determine if treatment inhibits the in-vitro cockroach antigen binding to B-cells after 6-months of treatment with cockroach SCIT, using the per protocol allergenic extract doses. This result is an indicator of immune modulation over time, however its clinical significance is unclear.
Time Frame: Baseline through 6-months of treatment
Population: Intent-to-treat
Measure: Mean (Standard Error); unit: Percent antibody binding
Arm/Group | Glycerinated German Cockroach Allergenic Extract
Number analyzed (Participants) | 10
Percent antibody binding | -42.8 (8.3)
Statistical Analysis 1: Comparison: Glycerinated German Cockroach Allergenic Extract; Test type: Superiority or Other; p < 0.0001, Change; Change = -42.8, 95% CI 2-sided [-59.4 to -26.2] — Numerator is geometric mean post-baseline FAB. Denominator is baseline FAB

ADVERSE EVENTS:
Groups:
- Experimental: German Cockroach Allergenic Extract: Participants received weekly escalating doses of glycerinated German cockroach allergenic extract administered via the subcutaneous route up to a Maximum Study Dose of 0.6 ml of extract at a concentration of 1:20 wt/vol.
Arm/Group | Experimental: German Cockroach Allergenic Extract
Serious Adverse Events (participants affected / at risk) | 2/10
Other Adverse Events (participants affected / at risk) | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental: German Cockroach Allergenic Extract (N=10)
Bronchitis (Infections and infestations) | 1 (1)
Localised infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental: German Cockroach Allergenic Extract (N=10)
Ear pruritus (Ear and labyrinth disorders) | 2 (4)
Eye pruritus (Eye disorders) | 1 (2)
Eye swelling (Eye disorders) | 1 (2)
Lacrimation increased (Eye disorders) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Lip pain (Gastrointestinal disorders) | 1 (1)
Lip swelling (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Influenza like illness (General disorders) | 1 (1)
Injection site anaesthesia (General disorders) | 1 (1)
Injection site eczema (General disorders) | 1 (1)
Injection site erosion (General disorders) | 2 (2)
Injection site erythema (General disorders) | 6 (15)
Injection site haemorrhage (General disorders) | 1 (1)
Injection site pain (General disorders) | 2 (4)
Injection site pruritus (General disorders) | 9 (53)
Injection site swelling (General disorders) | 9 (43)
Injection site urticaria (General disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1)
Blood urine present (Investigations) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (7)
Wisdom teeth removal (Surgical and medical procedures) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No